CLINICAL TRIAL: NCT06537362
Title: Comparative Evaluation of the Use of a Mouthpiece With Integrated Cheek Support vs. Manual Cheek Support During Respiratory Oscillometry Measurements
Brief Title: Mouthpiece With Integrated Cheek Support vs. Manual Cheek Support During Respiratory Oscillometry
Acronym: COMICUSROM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Raffaele Dellaca, professor, Politecnico di Milano
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CheekHolder
Record Dates: First submitted 2024-07-08; First posted 2024-08-05 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Morbidity; Lung Function Decreased
Keywords: Oscillometry
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): During oscillometry measures, the subject's cheeks are manually supported by an expert (Gold Standard method)
- Cheek Holder (Experimental): During oscillometry measures, the subject's cheeks are supported by an integrated cheek support in the mouthpiece
  Interventions: Device: Mouthpiece with cheek-holder

INTERVENTIONS:
Device: Mouthpiece with cheek-holder — A cheek support integrated into the mouthpiece is used for the measures
  Arms: Cheek Holder

SUMMARY:
The study aims to evaluate the measurement accuracy of respiratory impedance during oscillometry (or Forced Oscillation Technique - FOT) under the following conditions: 1)The subject's cheeks are manually supported by an expert (Gold Standard method), 2) The subject's cheeks are supported by an integrated cheek support in the mouthpiece.

It is a prospective, randomized, cross-over study on Subjects who will present themselves at the offices of the participating doctors, aged between 5 and 75 years. The primary outcome is to Compare the respiratory impedance measurements under the two measurement conditions. Secondary Objectives are to: i)evaluate the patient's comfort during the measurement with the cheek support and compare this comfort to the gold standard condition; ii) assess the maximum and minimum face dimensions of the recruited subjects that allow for effective and comfortable cheek support; iii) evaluate the type and frequency of measurement errors introduced by the use of the integrated cheek support in the mouthpiece.

DETAILED DESCRIPTION:
Study design: prospective, randomized, cross-over study. Study population: Subjects who will present themselves at the participating doctors' offices. Inclusion criteria: subjects aged between 5 and 75 years. Exclusion criteria: Subjects unable to follow the study procedures or with any physical or mental condition deemed unsuitable by the doctor will be excluded from the study.

Study protocol: the measurement protocol will consist of measuring the subject's facial morphological parameters and respiratory impedance parameters, followed by the administration of a questionnaire on perceived comfort. The procedure will be performed in a seated position.

Measurements:

1. Morphological Parameters Using a sliding caliper. The following anatomical distances will be measured on the seated subject, looking straight ahead with teeth together, facial muscles relaxed, and mouth closed: a) BIGONIAL WIDTH: The straight-line distance between the right and left angles of the mandible; b) LIP LENGTH: The straight-line distance between the right and left corners of the closed mouth."
2. Respiratory Impedance. The impedance measurement will be performed using the Resmon FIRST (Restech srl, Milan, Italy). Repeated measurements will be taken for each subject three times (TRIPLICATE) over 10 breaths with mono-frequency oscillations at 5 Hz. The enrolled subjects will perform the following measurements in a random order:

   * One TRIPLICATE session of respiratory impedance with cheeks supported by study personnel.
   * One TRIPLICATE session of respiratory impedance with cheeks supported by the cheek support. The study personnel will record any operator errors associated with preparing and using the cheek support on the enrolled participants.
3. Comfort Evaluation Questionnaire. At the end of the measurements, each participant will be asked to complete a comfort evaluation questionnaire regarding their experience during the procedure. Currently, no commercial devices are similar to the cheek support being tested. Therefore, the questionnaire is a modified version of a questionnaire previously used to evaluate the comfort of mechanical respirators worn on patients' faces during the coronavirus disease (COVID-19) period (Respirator Comfort, Wearing Experience, and Function Instrument (R-COMFI)3). The questionnaire aims to cover sensations of discomfort and general impressions of using the mouthpiece with cheek support during respiratory oscillometry measurements.

Sample size: The total number of subjects to be enrolled in the study is 55. This number was determined based on the following assumptions:

* Type-I error (α) = 5%, study power (1-β) >= 80%
* Uniform distribution of subjects in the following age groups: 6-17, 18-75 years
* Range of Resistance (Rrs) = 2...15 cmH2O/(L/s)
* Range of Reactance (Xrs) = 0...-14 cmH2O/(L/s)
* Minimum expected differences: the investigators set the minimum expected difference at 10% with a minimum value of 0.1 cmH2O/(L/s) (see table below)
* Expected standard deviation of variation: the investigators assume the expected standard deviation of variation to be the standard deviation of the short-term repeatability of oscillometry measurements reported in the literature (see table below)
* Dropout rate = 10%

Data analysis:

1. Comparison between the Cheek Holder Mouthpiece and Operator Support. The differences between the measurements taken with manual cheek support and those taken with the cheek holder will be analyzed. The two methods will be considered equivalent if the mean difference between the results and the 95% confidence interval of the Deming regression fall within the expected short-term variability of the technique for the tested population. Specifically:

   * For Rrs, a difference within 17% in adults and 27% in children, with a minimum acceptable difference of 1 cmH2O/(L/s), will be considered acceptable.
   * For Xrs, a difference within 37% in adults and 40% in children, with a minimum acceptable difference of 0.5 cmH2O/(L/s), will be considered acceptable.
2. Evaluation of Patient Comfort. The comfort of each patient will be assessed using a scoring system associated with specific questions. The total scores obtained with the two methodologies will be compared using a paired t-test or alternative tests for non-parametric distributions.
3. Evaluation of the Impact of Face Dimensions on FOT Test Accuracy. The impact of face dimensions on the effectiveness of the cheek holder support will be assessed by investigating the presence of a correlation between the differences in results obtained with the cheek holder and those obtained with manual support by the physician relative to lip length (LIP) and bigonial width. The type and frequency of user errors will be summarized for the entire population and for each age group using descriptive statistics (mean and standard deviation or median and ranges, as appropriate).

ELIGIBILITY:
Inclusion Criteria:

* subjects aged between 5 and 75 years

Exclusion Criteria:

* Subjects unable to follow the study procedures or with any physical or mental condition deemed unsuitable by the doctor will be excluded from the study

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
impedance measurements | within session (about 15 min)
  Compare the respiratory respiratory resistance (cmH2O*s/L) and reactance (cmH2O*s/L) at 5 Hz under the two measurement conditions

SECONDARY OUTCOMES:
evaluate patient's comfort during the measurement with the cheek support | within session (about 15 min)
  evaluate the patient's comfort during the measurement with the cheek support and compare this comfort to the gold standard condition as quantified by the questionnaire
face dimensions allowing for effective and comfortable cheek support | within session (about 15 min)
  assess the maximum and minimum face dimensions (to lip length and bigonial width) of the recruited subjects that allow for effective and comfortable cheek support as detailed in the Data Analysis section
evaluate the type and frequency of measurement errors | within session (about 15 min)
  evaluate the type and frequency of measurement errors introduced by the use of the integrated cheek support in the mouthpiece.

CONTACTS AND LOCATIONS:
Locations (1):
- Allergy and Pneumology Outpatient Clinic, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No